CLINICAL TRIAL: NCT01954056
Title: Hydrocortisone Treatment of Cardiovascular Insufficiency in Term and Late Preterm Infants: A Randomized Controlled Trial
Brief Title: Hydrocortisone for Term Hypotension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: NICHD Neonatal Research Network (Network)
Collaborators: National Center for Research Resources (NCRR) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NICHD-NRN-0052; U10HD021364 (NIH); U10HD040689 (NIH); U10HD021385 (NIH); U10HD027851 (NIH); U10HD027853 (NIH); U10HD027856 (NIH); U10HD027904 (NIH); U10HD027880 (NIH); U10HD034216 (NIH); U10HD021373 (NIH); U10HD040492 (NIH); U10HD053109 (NIH); U10HD040461 (NIH); U10HD068244 (NIH); U10HD068263 (NIH); U10HD068270 (NIH); U10HD068278 (NIH); U10HD068284 (NIH); U10HD036790 (NIH)
Record Dates: First submitted 2013-09-26; First posted 2013-10-01 (Estimated); Results first posted 2019-04-02 (Actual); Last update posted 2021-07-06 (Actual); Status verified 2021-07

CONDITIONS: Infant, Newborn, Diseases; Cardiovascular Insufficiency
Keywords: NICHD Neonatal Research Network; Mechanical ventilation; Intubation; Neurodevelopmental impairment
MeSH Terms: conditions — Infant, Newborn, Diseases | interventions — Hydrocortisone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hydrocortisone (Active Comparator): hydrocortisone (hydrocortisone sodium succinate, plain; will not have benzyl alcohol) given through intravenous line or by intramuscular injection if no intravenous line
  Interventions: Drug: Hydrocortisone
- Placebo (Placebo Comparator): Saline placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Hydrocortisone — • 7 day course of hydrocortisone (hydrocortisone sodium succinate, plain; will not have benzyl alcohol) given through intravenous line or by intramuscular injection if no intravenous line).
  1 mg/kg loading dose x 1; 0.5 mg/kg q 6 hours x 12 doses; 0.5 mg/kg q 12 hours x 4 doses; 0.5 mg/kg q day x 1 dose
  Arms: Hydrocortisone
Drug: Placebo — 7 days of intravenous or intramuscular placebo (normal saline in equal volume)
  1 mg/kg loading dose x 1; 0.5 mg/kg q 6 hours x 12 doses; 0.5 mg/kg q 12 hours x 4 doses; 0.5 mg/kg q day x 1 dose
  Arms: Placebo

SUMMARY:
This trial will evaluate the effects of a 7-day course of hydrocortisone therapy on short-term morbidity, cardiovascular function, long-term neurodevelopment, and mortality in critically ill, term and late preterm infants diagnosed with cardiovascular insufficiency as defined by a need for inotrope therapy in the first 72 hours of age.

DETAILED DESCRIPTION:
Cardiovascular insufficiency is common and potentially life-threatening in critically ill term and late preterm newborns admitted to the newborn intensive care unit (NICU) in the first few days of age.

This study proposes to conduct a multicenter, randomized, masked, placebo-controlled trial within the Neonatal Research Network (NRN). This trial will evaluate the effects of a 7-day course of hydrocortisone therapy on short-term morbidity, cardiovascular function, long-term neurodevelopment, and mortality in critically ill, term and late preterm infants diagnosed with cardiovascular insufficiency as defined by a need for inotrope therapy in the first 72 hours of age.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age greater than or equal to 34 weeks at birth
* Admitted to the center NICU by 48 hours of age
* Intubated and mechanically ventilated for a minimum of 2 hours before 72 hours postnatal age

Exclusion Criteria:

* Receiving ECMO
* Intubated for the sole purpose of anticipated surgery or airway anomalies
* Treatment will be limited based on poor prognosis
* Receiving dexamethasone or hydrocortisone
* Receiving ibuprofen or indomethacin
* Congenital heart disease
* Hypotension thought to result from specific, immediately remediable factors including placental hemorrhage, acute hemorrhage or tension pneumothorax
* Pituitary hypoplasia or congenital adrenal hyperplasia
* Any chromosomal disorder
* Hypertension in the absence of inotrope therapy as defined by mean arterial blood pressure > 95th percentile
* Initiation of whole body cooling for moderate or severe neonatal encephalopathy
* Brain disorders or any other known structural abnormality
* Major anomalies

Min Age: 34 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2014-06-19 (Actual); Primary Completion 2018-03-20 (Actual); Study Completion 2018-03-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michele C Walsh, MD, Principal Investigator — Case Western Reserve University, Rainbow Babies and Children's Hospital; Seetha Shankaran, MD, Principal Investigator — Wayne State University; Abbot R Laptook, MD, Principal Investigator — Brown University, Women & Infants Hospital of Rhode Island; Ron N Goldberg, MD, Principal Investigator — Duke University; Barbara J Stoll, MD, Principal Investigator — Emory University; Brenda B Poindexter, MD, MS, Principal Investigator — Indiana University; Abhik Das, PhD, Principal Investigator — RTI International; Krisa P Van Meurs, MD, Principal Investigator — Stanford University; Kurt Schibler, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati; Waldemar Carlo, MD, Principal Investigator — University of Alabama at Birmingham; Edward F Bell, MD, Principal Investigator — Michele C Walsh, MD Study Principal Investigator Case Western Reserve University, Rainbow Babies and Children's Hospital Seetha Shankaran, MD Study Principal Investigator Wayne State University Abbot R Laptook, MD Study Principal Investigator Brown Un; Erika Fernandez, MD, Study Chair — University of New Mexico; Myra Wycoff, MD, Principal Investigator — University of Texas, Southwestern Medical Center at Dallas; Kathleen A Kennedy, MD, MPH, Principal Investigator — The University of Texas Health Science Center, Houston; Barbara Schmidt, MD, Principal Investigator — University of Pennsylvania; Carl T D'Angio, MD, Principal Investigator — University of Rochester; Uday Devaskar, MD, Principal Investigator — University of California, Los Angeles; Leif Nelin, MD, Principal Investigator — Research Institute at Nationwide Children's Hospital; William Truog, MD, Principal Investigator — Children's Mercy Hospital Kansas City
Locations (18):
- United States (18):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of California - Los Angeles, Los Angeles, California
  - Stanford University, Palo Alto, California
  - Emory University, Atlanta, Georgia
  - Indiana University, Indianapolis, Indiana
  - University of Iowa, Iowa City, Iowa
  - Wayne State University, Detroit, Michigan
  - Children's Mercy Hospital, Kansas City, Missouri
  - University of New Mexico, Albuquerque, New Mexico
  - University of Rochester, Rochester, New York
  - RTI International, Durham, North Carolina
  - Duke University, Durham, North Carolina
  - Cincinnati Children's Medical Center, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - Research Institute at Nationwide Children's Hospital, Columbus, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Texas Southwestern Medical Center at Dallas, Dallas, Texas
  - University of Texas Health Science Center at Houston, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: NICHD Neonatal Research Network site — http://neonatal.rti.org/
- See also: NICHD Pregnancy & Perinatology Branch — http://www.nichd.nih.gov/about/org/der/branches/ppb/Pages/overview.aspx

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Infants < 48 hours of age and born at ≥ 34 weeks gestational age were screened for the study between June 2014 and July 2015 at the 16 NRN Clinical Centers. Those who were intubated and on mechanical ventilation for at least 2 hours within the first 72 hours were considered for the study.
Groups:
- Hydrocortisone: hydrocortisone (hydrocortisone sodium succinate, plain; will not have benzyl alcohol) given through intravenous line or by intramuscular injection if no intravenous line
  Hydrocortisone: • 7 day course of hydrocortisone (hydrocortisone sodium succinate, plain; will not have benzyl alcohol) given through intravenous line or by intramuscular injection if no intravenous line).
  1 mg/kg loading dose x 1; 0.5 mg/kg q 6 hours x 12 doses; 0.5 mg/kg q 12 hours x 4 doses; 0.5 mg/kg q day x 1 dose
- Placebo: Saline placebo
  Placebo: 7 days of intravenous or intramuscular placebo (normal saline in equal volume)
  1 mg/kg loading dose x 1; 0.5 mg/kg q 6 hours x 12 doses; 0.5 mg/kg q 12 hours x 4 doses; 0.5 mg/kg q day x 1 dose
Period: Birth to 60 Days of Life
Arm/Group | Hydrocortisone | Placebo
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0
Period: Birth to 22-26 Mos. Corrected GA
Arm/Group | Hydrocortisone | Placebo
Started | 6 | 6
Completed | 5 | 6
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Hydrocortisone: Hydrocortisone: 7 day course of hydrocortisone (hydrocortisone sodium succinate, plain; will not have benzyl alcohol) given through intravenous line or by intramuscular injection if no intravenous line).
  1 mg/kg loading dose x 1; 0.5 mg/kg q 6 hours x 12 doses; 0.5 mg/kg q 12 hours x 4 doses; 0.5 mg/kg q day x 1 dose
- Placebo: Saline placebo: 7 days of intravenous or intramuscular placebo (normal saline in equal volume)
  1 mg/kg loading dose x 1; 0.5 mg/kg q 6 hours x 12 doses; 0.5 mg/kg q 12 hours x 4 doses; 0.5 mg/kg q day x 1 dose
- Total: Total of all reporting groups
Arm/Group | Hydrocortisone | Placebo | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Continuous [Mean (Standard Deviation); unit: weeks] — Age refers to the infant and is measured as gestational age in weeks.
  weeks | 37.5 (2.2) | 39.4 (1.8) | 38.4 (2.2)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 4 | 2 | 6
  Female | 2 | 4 | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 3 | 5 | 8
  Unknown or Not Reported | 2 | 0 | 2
Maternal Race [Count of Participants; unit: Participants]
  Black | 3 | 2 | 5
  White | 3 | 2 | 5
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 1 | 1
Maternal Age, Continuous [Mean (Standard Deviation); unit: years] | 32.2 (7.6) | 26.7 (9.5) | 29.4 (8.7)
Birth weight [Mean (Standard Deviation); unit: grams] | 3415 (669.3) | 3120.3 (541) | 3267.7 (600.3)
Length [Mean (Standard Deviation); unit: cm] | 50.1 (2.3) | 49.8 (1.5) | 49.9 (1.9)
Head circumference [Mean (Standard Deviation); unit: cm] | 34.4 (2) | 34.5 (3.5) | 34.5 (2.7)
Apgar score less than 3 at 1 minute [Count of Participants; unit: Participants] — The Apgar score is determined by evaluating the newborn baby on five simple criteria on a scale from zero to two, then summing up the five values thus obtained. Total Apgar scores range from 0 to 10. This measure is calculated at 1 minute after birth as Yes if total Apgar is less than 3. No, otherwise.
  Participants
    No | 2 | 4 | 6
    Yes | 4 | 2 | 6
Apgar score less than 3 at 5 minutes [Count of Participants; unit: Participants] — The Apgar score is determined by evaluating the newborn baby on five simple criteria on a scale from zero to two, then summing up the five values thus obtained. Total Apgar scores range from 0 to 10. This measure is calculated at 5 minutes after birth as Yes if total Apgar is less than 3. No, otherwise.
  Participants
    No | 5 | 6 | 11
    Yes | 1 | 0 | 1
Apgar score less than 3 at 10 minutes [Count of Participants; unit: Participants] — The Apgar score is determined by evaluating the newborn baby on five simple criteria on a scale from zero to two, then summing up the five values thus obtained. Total Apgar scores range from 0 to 10. This measure is calculated at 10 minutes after birth as Yes if total Apgar is less than 3. No, otherwise.
  Participants
    No | 3 | 3 | 6
    Yes | 0 | 0 | 0
    Unknown | 3 | 3 | 6
Infant Outborn [Count of Participants; unit: Participants]
  No | 4 | 2 | 6
  Yes | 2 | 4 | 6
Oxygen [Count of Participants; unit: Participants] — Collected during Resuscitation at Delivery
  Participants
    Yes | 6 | 6 | 12
    No | 0 | 0 | 0
Bagging and Mask [Count of Participants; unit: Participants] — Collected during Resuscitation at Delivery
  Participants
    No | 1 | 2 | 3
    Yes | 5 | 4 | 9
Chest Compression [Count of Participants; unit: Participants] — Collected during Resuscitation at Delivery
  Participants
    No | 5 | 5 | 10
    Yes | 1 | 1 | 2
Intubation [Count of Participants; unit: Participants] — Collected during Resuscitation at Delivery
  Participants
    No | 4 | 1 | 5
    Yes | 2 | 5 | 7
Medications or volume expanders [Count of Participants; unit: Participants] — Collected during Resuscitation at Delivery
  Participants
    No | 5 | 3 | 8
    Yes | 1 | 3 | 4
Maternal marital Status [Count of Participants; unit: Participants]
  Married | 1 | 1 | 2
  Single | 5 | 5 | 10
Maternal gravida [Median (Full Range); unit: Number of pregnancies] — The number of confirmed pregnancies.
  Number of pregnancies | 2.5 [1 to 6] | 1 [1 to 7] | 2 [1 to 7]
Maternal parity [Median (Full Range); unit: Number of successful pregnancies] — The number of pregnancies reaching 20 weeks and 0 days of gestation or beyond, regardless of the number of fetuses or outcomes, including this delivery.
  Number of successful pregnancies | 2.5 [1 to 4] | 1 [1 to 4] | 2 [1 to 4]
Maternal multiple birth [Count of Participants; unit: Participants]
  No | 6 | 6 | 12
  Yes | 0 | 0 | 0
Maternal prenatal care [Count of Participants; unit: Participants]
  No | 2 | 1 | 3
  Yes | 4 | 5 | 9
Maternal antenatal steroids [Count of Participants; unit: Participants]
  No | 6 | 6 | 12
  Yes | 0 | 0 | 0
Maternal documented chorioamnionitis [Count of Participants; unit: Participants]
  No | 5 | 6 | 11
  Yes | 1 | 0 | 1
Placental pathology performed [Count of Participants; unit: Participants]
  No | 1 | 1 | 2
  Yes | 2 | 3 | 5
  Unknown | 3 | 2 | 5
Final mode of delivery [Count of Participants; unit: Participants]
  Vaginal vertex | 3 | 2 | 5
  Cesarean section | 3 | 3 | 6
  Unknown | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Death
Description: This is measured as Yes if an infant died between birth and 22-26 months corrected gestational age; Otherwise, No.
Time Frame: Birth to 22-26 months corrected gestational age
Population: The analysis population includes all randomized infants recruited from critically ill, term and late preterm infants diagnosed with cardiovascular insufficiency as defined by a need for inotrope therapy in the first 72 hours of age.
Measure: Count of Participants; unit: Participants
Arm/Group | Hydrocortisone | Placebo
Number analyzed (Participants) | 6 | 6
Participants
  No | 6 | 6
  Yes | 0 | 0

2. Primary Outcome: Number of Participants With Neurodevelopmental Impairment
Description: This is measured as Yes if an any hearing impairment or visual impairment is noted, if non-normal gross motor function level is noted, any seizures have been noted, or if the cognitive, language, or motor scores of the Bayley III score are more than 1 standard deviation below the average; Otherwise, No.
Time Frame: Birth to 22-26 months corrected gestational age
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Hydrocortisone | Placebo
Number analyzed (Participants) | 6 | 6
Participants
  Yes | 3 | 3
  No | 3 | 3

3. Primary Outcome: Number of Participants With Death or Neurodevelopmental Impairment
Description: A composite outcome that measures the occurrence of death or neurodevelomental impairment between birth and 22-26 months corrected gestational age.
Time Frame: Birth to 22-26 months corrected gestational age
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Hydrocortisone | Placebo
Number analyzed (Participants) | 6 | 6
Participants
  Yes | 3 | 3
  No | 3 | 3

4. Secondary Outcome: Duration of Mechanical Ventilation
Description: This is measured as the number of days between birth and 60 days of life of mechanical ventialtion of laryngeal intubation.
Time Frame: Birth to 60 days of life
Population: as for outcome 1
Measure: Median (Full Range); unit: Days
Arm/Group | Hydrocortisone | Placebo
Number analyzed (Participants) | 6 | 6
Days | 8 [3 to 10] | 11 [3 to 19]

5. Secondary Outcome: Days to Full Feeds
Description: The day of life at which full nipple feeds were reached between birth and 60 days of life. Full nipple feeds are defined as at least 120 mg/kg/day.
Time Frame: Birth to 60 days of life
Population: The analysis population includes all randomized infants recruited from critically ill, term and late preterm infants diagnosed with cardiovascular insufficiency as defined by a need for inotrope therapy in the first 72 hours of age. Excludes 4 infants (Hydrocortisone: 1, Placebo: 3) without information on full feeds.
Measure: Median (Full Range); unit: Days
Arm/Group | Hydrocortisone | Placebo
Number analyzed (Participants) | 5 | 3
Days | 16 [12 to 23] | 18 [8 to 22]

6. Secondary Outcome: Number of Participants With Need for Gastronomy Tube
Description: This is measured as Yes if a gastronomy tube was placed anytime prior to final status between birth and 60 days of life; Otherwise, No
Time Frame: Birth to 60 days of life
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Hydrocortisone | Placebo
Number analyzed (Participants) | 6 | 6
Participants
  No | 6 | 6
  Yes | 0 | 0

7. Secondary Outcome: Duration of Oxygen Requirement
Description: This is measured as the number of days between birth and 60 days of life that an infant was on oxygen in the hospital.
Time Frame: Birth to 60 days of life
Population: as for outcome 1
Measure: Median (Full Range); unit: Days
Arm/Group | Hydrocortisone | Placebo
Number analyzed (Participants) | 6 | 6
Days | 15.5 [3 to 33] | 18 [5 to 25]

8. Secondary Outcome: Number of Participants With Need for Home Oxygen
Description: This is measured as Yes if an infant was discharged to home while on oxygen between birth and 60 days of life; Otherwise, No.
Time Frame: Birth to 60 days of life
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Hydrocortisone | Placebo
Number analyzed (Participants) | 5 | 6
Participants
  No | 5 | 4
  Yes | 0 | 2

9. Secondary Outcome: Hospital Length of Stay
Description: This is measured as the number of days between birth and 60 days of life that an infant was in the hospital. Infants who died or transferred to another care facility were not included.
Time Frame: Birth to 60 days of life
Population: as for outcome 1
Measure: Median (Full Range); unit: Days
Arm/Group | Hydrocortisone | Placebo
Number analyzed (Participants) | 5 | 5
Days | 27 [14 to 60] | 24 [14 to 38]

10. Secondary Outcome: Number of Participants With Renal Insufficiency
Description: This is measured as Yes if an infant had renal insufficieny between birth and 60 days of life; Otherwise, No. Renal insufficiency is defined as creatinine less than 2 during 7 days after first treatment
Time Frame: Birth to 60 days of life
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Hydrocortisone | Placebo
Number analyzed (Participants) | 6 | 6
Participants
  No | 6 | 6
  Yes | 0 | 0

11. Secondary Outcome: Number of Participants With Necrotizing Enterocolitis
Description: This is measured as Yes if an infant necrotizing enterocolitis (NEC) between birth and 60 days of life; Otherwise, No. NEC could be proven with or without surgery
Time Frame: Birth to 60 days of life
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Hydrocortisone | Placebo
Number analyzed (Participants) | 6 | 6
Participants
  No | 5 | 6
  Yes | 1 | 0

12. Secondary Outcome: Number of Participants With Need for ECMO Therapy
Description: This is measured as Yes if an infant received ECMO treatment anytime between birth and 60 days of life; Otherwise, No. Extracorporeal membrane oxygenation (ECMO) is a treatment that uses a pump to circulate blood through an artificial lung back into the bloodstream of a very ill baby.
Time Frame: Birth to 60 days of life
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Hydrocortisone | Placebo
Number analyzed (Participants) | 6 | 6
Participants
  No | 6 | 6
  Yes | 0 | 0

13. Secondary Outcome: Number of Participants With Inotrope Exposure
Description: This is measured as Yes if an infant was receiving inotropes on the specific day after the initiation of study drug.
Time Frame: 24 hours prior to study drug administration through 3 days post study drug administration.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Hydrocortisone | Placebo
Number analyzed (Participants) | 6 | 6
Participants
  Day 3: No | 4 | 4
  Day 3: Yes | 2 | 2
  Day 5: No | 5 | 4
  Day 5: Yes | 1 | 2
  Day 7: No | 5 | 5
  Day 7: Yes | 1 | 1

14. Secondary Outcome: Inotrope Duration
Description: This is calculated as the number of days on inotropes starting 24 hours prior to initiation of study drug, during the 7-day study drug administration period, and for 3 days after the study drug.
Time Frame: 24 hours prior to study drug administration through 3 days post study drug administration.
Population: as for outcome 1
Measure: Median (Full Range); unit: days
Arm/Group | Hydrocortisone | Placebo
Number analyzed (Participants) | 6 | 6
days | 3 [1 to 8] | 3 [1 to 8]

15. Secondary Outcome: Maximum Inotrope Dose
Description: This is calculated as the maximum dose of all inotropes in the 10 days following the initiation of study drug administration. For the purposes of this calculation, dopamine and dobutamine doses were considered equivalent and 0.01 mcg/kg/min of epinephrine was equal to 5 mcg/kg/min of dopamine.
Time Frame: From start of study drug administration (7 days) through 3 days post study drug administration.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mcg/kg/min
Arm/Group | Hydrocortisone | Placebo
Number analyzed (Participants) | 6 | 6
mcg/kg/min | 9.5 (2.9) | 14.7 (12.6)

16. Secondary Outcome: Oxygenation Index
Description: This is calculated as fraction of inspired oxygen (FiO2), as a percentage, multiplied by the mean airway pressure divided by partial pressure of oxygen in arterial blood (PaO2), during study drug administration. A lower oxygenation index is better.
Time Frame: Birth to 60 days of life
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Oxygenation Index
Arm/Group | Hydrocortisone | Placebo
Number analyzed (Participants) | 6 | 6
Oxygenation Index
  Before dose 1 | 10.7 (6.1) | 14.5 (8.6)
  Before dose 5: number analyzed (Participants) | 6 | 5
  Before dose 5 | 7 (3.7) | 14.9 (6.9)
  Before dose 9: number analyzed (Participants) | 5 | 5
  Before dose 9 | 6.6 (2.1) | 10.4 (5.3)
  Before dose 13: number analyzed (Participants) | 5 | 5
  Before dose 13 | 5.8 (3) | 9.2 (4.2)
  Before dose 15: number analyzed (Participants) | 3 | 3
  Before dose 15 | 4.7 (2) | 9.3 (0.8)
  Before dose 17: number analyzed (Participants) | 3 | 3
  Before dose 17 | 5.9 (3.2) | 7.9 (1.1)
  Before dose 18: number analyzed (Participants) | 1 | 3
  Before dose 18 | 3.7 | 9.1 (4.6)

17. Secondary Outcome: Respiratory Severity
Description: This is calculated as fraction of inspired oxygen (FiO2), as a percentage, multiplied by the mean airway pressure during study drug administration. Higher score means more severe.
Time Frame: Birth to 60 days of life
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage of inspired oxygen * cmH2O
Arm/Group | Hydrocortisone | Placebo
Number analyzed (Participants) | 6 | 6
Percentage of inspired oxygen * cmH2O
  Before dose 1 | 726.8 (371) | 1184.7 (518.7)
  Before dose 5: number analyzed (Participants) | 6 | 5
  Before dose 5 | 518.8 (272.5) | 1041.2 (432.6)
  Before dose 9: number analyzed (Participants) | 5 | 5
  Before dose 9 | 531.6 (196.5) | 925.8 (611.8)
  Before dose 13: number analyzed (Participants) | 5 | 5
  Before dose 13 | 414.6 (230) | 776.8 (411.2)
  Before dose 15: number analyzed (Participants) | 4 | 3
  Before dose 15 | 423 (158.8) | 899 (453.4)
  Before dose 17: number analyzed (Participants) | 3 | 4
  Before dose 17 | 323 (117.8) | 785.8 (463.2)
  Before dose 18: number analyzed (Participants) | 2 | 3
  Before dose 18 | 308.5 (139.3) | 694.7 (274)

18. Secondary Outcome: Number of Participants With Fluid Boluses Given
Description: This is measured as Yes if an infant received fluid boluses anytime before or during study drug administration between birth and 60 days of life; Otherwise, No.
Time Frame: Birth to 60 days of life
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Hydrocortisone | Placebo
Number analyzed (Participants) | 6 | 6
Participants
  Before dose 1: No | 2 | 2
  Before dose 1: Yes | 4 | 4
  Before dose 5: No | 5 | 4
  Before dose 5: Yes | 1 | 2
  Before dose 9: No | 5 | 5
  Before dose 9: Yes | 1 | 1
  Before dose 13: No | 5 | 6
  Before dose 13: Yes | 1 | 0
  Before dose 15: number analyzed (Participants) | 6 | 5
  Before dose 15: No | 6 | 4
  Before dose 15: Yes | 0 | 1
  Before dose 17: No | 6 | 6
  Before dose 17: Yes | 0 | 0
  Before dose 18: No | 6 | 6
  Before dose 18: Yes | 0 | 0

19. Secondary Outcome: Number of Boluses Given
Description: The number of fluid boluses given per participant, if any, before or during study drug administration between birth and 60 days of life
Time Frame: Birth to 60 days of life
Population: as for outcome 1
Measure: Median (Full Range); unit: Boluses
Arm/Group | Hydrocortisone | Placebo
Number analyzed (Participants) | 5 | 5
Boluses
  Before dose 1: number analyzed (Participants) | 4 | 4
  Before dose 1 | 3 [1 to 7] | 3 [2 to 8]
  Before dose 5: number analyzed (Participants) | 1 | 2
  Before dose 5 | 2 [2 to 2] | 1 [1 to 1]
  Before dose 9: number analyzed (Participants) | 1 | 1
  Before dose 9 | 2 [2 to 2] | 1 [1 to 1]
  Before dose 13: number analyzed (Participants) | 1 | 0
  Before dose 13 | 1 [1 to 1] |
  Before dose 15: number analyzed (Participants) | 0 | 1
  Before dose 15 |  | 1 [1 to 1]

ADVERSE EVENTS:
Time Frame: 10 days
Arm/Group | Hydrocortisone | Placebo
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 1/6 | 0/6
Other Adverse Events (participants affected / at risk) | 0/6 | 1/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hydrocortisone (N=6) | Placebo (N=6)
HYPERBILIRUBINEMIA REQUIRING EXCHANGE TRANSFUSION (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
HYPERTENSION, NEW AND SUSTAINED (Cardiac disorders) | 1 (2) | 0 (0)
ADRENAL INSUFFICIENCY (Endocrine disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hydrocortisone (N=6) | Placebo (N=6)
ATRIAL TACHYCARDIA (Cardiac disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
The study was closed to enrollment after 12 participants due to slow recruitment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigators must adhere to the Neonatal Research Network Publication policies

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-04-02): https://cdn.clinicaltrials.gov/large-docs/56/NCT01954056/Prot_SAP_000.pdf